CLINICAL TRIAL: NCT03115138
Title: Evaluation of Circulating Tumor DNA as a Theranostic Marker in the Management of Glioblastomas.
Acronym: Bi-GLAM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator choice
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2015_843_0029
Record Dates: First submitted 2017-04-04; First posted 2017-04-14 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Glioblastoma; Molecular Disease
Keywords: Biopsy
MeSH Terms: conditions — Glioblastoma; Genetic Diseases, Inborn | interventions — Circulating Tumor DNA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with glial tumor (Other)
  Interventions: Other: Correlation between molecular anomalies of the primary tumor and circulating tumor DNA

INTERVENTIONS:
Other: Correlation between molecular anomalies of the primary tumor and circulating tumor DNA — The presence of a specific abnormality initially identified on the primary tumor and which can be quantified in the cDNA during the management will allow a better follow-up of the patient.

SUMMARY:
Glioblastomas (GBM) are rare tumors of poor prognosis and their treatment is based on surgery followed by radiochemotherapy. Clinical and imaging evaluation is not always straightforward: the more or less complete surgery, the pseudo-progression after radiochemotherapy, the radionecrosis, the diagnosis of the relapse and the follow-up under anti-angiogenic can pose problems Clinicians and radiologists. Accessibility to a plasma tumor molecular marker would greatly facilitate the follow-up of these patients.

It is now established for many cancers that circulating tumor DNA (cTNA) has the same molecular abnormalities as those identified in the primary tumor cells. Numerous studies have shown the prognostic value and diagnosis of the exploration of cDNA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with grade IV glial tumor (glioblastoma according to WHO criteria) for which an indication of surgical excision with radiochemotherapy was chosen at a specialized multidisciplinary meeting of neuro-oncology at the CHU Amiens-Picardy.
* Patients should:

  * be able to be followed at the CHU of Amiens throughout their treatment,
  * be at least 18 years of age,
  * be informed (or trusted) of the conditions and objectives of the study,
  * having given their free and informed consent in writing,
  * have a life expectancy of more than 6 months,
  * be affiliated to a social security scheme.

Exclusion Criteria:

* Patients with recurrent tumors.
* Patients supported for another histology.
* Medical, psychological or social conditions that do not allow for proper understanding of the procedures inherent in the study.
* Patients under tutelage, curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Presence of a correlation between the molecular abnormalities of the primary tumor and the circulating tumor DNA | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France